CLINICAL TRIAL: NCT05081349
Title: Treatment With Hydoxycarbamide and L-Carnitine in Adult Patients With Severe Forms of Sickle Cell Anemia: An Overview
Brief Title: Hydoxycarbamide and L-Carnitine Therapy in Sickle Cell Anemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa AA Khaled, Clinical Professor, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKhaled2021
Record Dates: First submitted 2021-09-24; First posted 2021-10-18 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2016-12

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea; Carnitine

STUDY DESIGN:
Intervention Model Description: Non-randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Hydra+L-Carnitine (Experimental): Hydroxycarbamide+ L-Carnitine+supportive treatment
  Interventions: Drug: Hydroxycarbamide 500 Mg Oral Capsule+L-Carnitine
- Hydra only (Active Comparator): Hydroxycarbamide+ supportive treatment
  Interventions: Drug: Hydroxycarbamide 500 Mg Oral Capsule
- L-Carnitine only (Active Comparator): L-Carnitine+ supportive treatment
  Interventions: Drug: L-Carnitine, 250 Mg Oral Capsule
- Supportive measures (No Intervention): Supportive only

INTERVENTIONS:
Drug: Hydroxycarbamide 500 Mg Oral Capsule+L-Carnitine — Combination therapy
  Other Names: Hydroxyurea+LC
  Arms: Hydra+L-Carnitine
Drug: Hydroxycarbamide 500 Mg Oral Capsule — Single agent
  Other Names: Hydroxyurea
  Arms: Hydra only
Drug: L-Carnitine, 250 Mg Oral Capsule — single agent
  Other Names: L-Carnitine
  Arms: L-Carnitine only

SUMMARY:
The role of the combination therapy of hydroxyurea and L-Carnitine was studied in thalassemic patients. nevertheless its role in sickle cell anemia patients was not investigated

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is a common monogenic disorder affecting over 100,000 people in the United States alone, and millions more worldwide. This often devastating disease is characterized by red blood cell (RBC) sickling; chronic hemolytic anemia; episodic vaso-occlusion associated with severe pain and inflammation; acute and cumulative organ damage that manifests as stroke, acute chest syndrome, sickle lung disease, pulmonary hypertension nephropathy and end-stage renal disease; and other chronic morbidities.

Lives of patients with SCD are characterized by frequent episodes of severe pain (vaso-occlusive events or "crises"); acute organ dysfunction, including a pneumonia-like syndrome termed acute chest syndrome, and strokes starting in childhood; and progressive multi-organ damage. Not surprisingly, patients with SCD have very high health care utilization (over $1 billion/year in healthcare costs in the United States alone, and a median life-expectancy of only ~45-58 years, compared to the life expectancy of 78.2 years overall in the United States.

Although it is licensed in the United States for administration to sickle cell patients who have ≥ 3 crises a year in steady state, hydroxyurea (HU) remains unlicensed in most countries where it is regarded as an experimental drug In those areas, where HU is unlicensed for SCD, it is offered to patients who have ≥ 5 crises a year; or 3-4 crises a year with either neutrophil count ≥ 10 × 109/L or platelet count ≥ 500 × 109/L in steady state ; bearing in mind that the reference range for neutrophil count in black people is 1-3 × 109/L, and is 100-300 × 109/L for platelets .

Since high neutrophil count in steady state is a marker of severe SCD , these criteria usually identify individuals who have a clinical course sufficiently severe to ensure that the benefits of hydroxyurea therapy justify the potential risks. HU therapy is offered if the patient does not want to have (more) children, and is weighed against any severe impairment of liver or kidney function, or blood cytopenia. HU is unlicensed in most countries because the long-term adverse effects are unknown, not because the clinical efficacy is in doubt. In fact, after over 9 years of follow-up, HbSS subjects who received HU in the US placebo-controlled trial, had significantly less painful crises, acute chest syndrome, and mortality . Potential long-term toxic effects that reduce enthusiasm for HU include teratogenicity, carcinogenesis and, for young children, impaired cognitive development.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sickle cell disease
* Not welling for pregnancy in females or to father a baby in males
* Frequent episodes
* Non-compliance to transfusion

Exclusion Criteria:

* <18 years
* Hypersensitivity to hydroxycarbamide or L-Carnitine
* Pregnancy
* Other chronic infection or inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
Hematological(HR) | 2-3 months
  Change of hemoglobin
Hematological response | 2-3 months
  Change of hematocrit

SECONDARY OUTCOMES:
Frequency of painful episodes/ blood transfusions | 1-year
  Change of frequency of painful episodes and blood transfusion

OTHER OUTCOMES:
Delayed effects | 12-18 months
  effect on long term complications as cardiovascular and cerebrovascular ones

CONTACTS AND LOCATIONS:
Overall Officials: Israa EM Ashry, Prof, Study Director — Assiut University- Faculty of Medicine
Locations (1):
- Safaa A A Khaled, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bunn HF. Pathogenesis and treatment of sickle cell disease. N Engl J Med. 1997 Sep 11;337(11):762-9. doi: 10.1056/NEJM199709113371107. No abstract available. PMID 9287233
- [Background] Rees DC, Williams TN, Gladwin MT. Sickle-cell disease. Lancet. 2010 Dec 11;376(9757):2018-31. doi: 10.1016/S0140-6736(10)61029-X. Epub 2010 Dec 3. PMID 21131035
- [Background] Platt OS, Brambilla DJ, Rosse WF, Milner PF, Castro O, Steinberg MH, Klug PP. Mortality in sickle cell disease. Life expectancy and risk factors for early death. N Engl J Med. 1994 Jun 9;330(23):1639-44. doi: 10.1056/NEJM199406093302303. PMID 7993409
- [Background] Kauf TL, Coates TD, Huazhi L, Mody-Patel N, Hartzema AG. The cost of health care for children and adults with sickle cell disease. Am J Hematol. 2009 Jun;84(6):323-7. doi: 10.1002/ajh.21408. PMID 19358302
- [Background] Elmariah H, Garrett ME, De Castro LM, Jonassaint JC, Ataga KI, Eckman JR, Ashley-Koch AE, Telen MJ. Factors associated with survival in a contemporary adult sickle cell disease cohort. Am J Hematol. 2014 May;89(5):530-5. doi: 10.1002/ajh.23683. Epub 2014 Feb 21. PMID 24478166